CLINICAL TRIAL: NCT01699607
Title: Test-retest Reproducibility of [11C]PHNO PET Using the Constant Infusion
Brief Title: Test-retest Reproducibility of [11C]PHNO PET Using the Constant Infusion Paradigm
Acronym: phno_amth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0910005822; R25MH071584 (NIH); 1P50CA196530-01 (NIH)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Nicotine Dependence; Healthy
Keywords: Cigarette Smokers; Healthy Non Smokers; Amphetamine; PET; Controls
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Amphetamine; Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- amphetamine (Experimental): There is only one arm to the study. All subjects will receive amphetamine at 0.5mg/kg prior to the second PET scan.
  Interventions: Drug: Amphetamine

INTERVENTIONS:
Drug: Amphetamine — All subjects will receive amphetamine to induce elevated dopamine levels in the brain at 0.5mg/kg
  Other Names: dextro-amphetamine

SUMMARY:
A research study designed to examine amphetamine-induced dopamine release using the PET imaging agent [11C]PHNO in tobacco smokers while currently smoking and during acute withdrawal and in nonsmokers. Twenty healthy men and women tobacco smokers and twenty healthy nonsmokers will be recruited. Each subject will participate in 1 MRI and up to 2 [11C]PHNO PET scans. On the study day subjects will participate in two [11C]PHNO scans (ideally, the two PET scans will be carried out in the same day). Three hours before the second PET scan, amphetamine (0.5 mg/kg, PO) will be administered. In smokers, the scan will occur at 10-21 days of smoking abstinence.

DETAILED DESCRIPTION:
To determine amphetamine-induced DA release in tobacco smokers while currently smoking and during acute withdrawal and in nonsmokers. Twenty healthy men and women tobacco smokers and twenty healthy nonsmokers will be recruited. Each subject will participate in 1 MRI and up to 2 [11C]PHNO PET scans. On the PET study day subjects will participate in two [11C]PHNO scans (ideally, the two PET scans will be carried out in the same day). Three hours before the second PET scan, amphetamine (0.5 mg/kg, PO) will be administered. In smokers, the set of scans will occur at 10-21 days of smoking abstinence. Smoking abstinence will be determined by carbon monoxide and urine cotinine (a breakdown product of nicotine in cigarette smoke) levels. Subjects will be asked to breathe into a breathalyzer to measure carbon monoxide and to provide a urine sample to measure cotinine. Smoking abstinence will be confirmed by carbon monoxide and cotinine levels that are reduced as compared to actively smoking. We hypothesize that smokers at 10-21 days of withdrawal will have amphetamine-induced DA release that is blunted compared to healthy nonsmokers.

Magnetic resonance imaging (MRI) scans (3 T) will be collected in each subject to co-register PET and MRI for image analysis. Within two weeks of the PET study, an MRI will be acquired at the Yale University MRI Center. Subjects will be taken through a ferromagnetic metal detector before entering the scan room. The acquisition sequence is a 3D fast spoiled grass (FSPGR) MR pulse sequence with an IR prep of 300 ms. (TE= 3.3 ms, flip angle=17 degrees; slice thickness= 1.2 mm) optimized for delineating gray matter/white matter/CSF boundaries. The small voxel size (0.93 X 1.2 X 0.93 mm) provides high-resolution volumetric images. MR images provide a matching anatomical atlas for creating individualized region-of-interest templates for each subject.

Subject preparation consists of two intravenous (IV) catheterizations and immobilization of the head. PET scans are acquired as subjects rest using an HRRT PET scanner (207 slices, resolution better than 3 mm FWHM). This resolution permits visualization of the PHNO and raclopride uptake in the ventral/dorsal striatum, in globus pallidus (GP) and substantia nigra (SN). A transmission scan using an orbiting 137Cs point-source is obtained for each emission scan. Motion correction will be performed dynamically with measurements from the Vicra (NDI Systems, Waterloo, Ontario) used by a dedicated list-mode reconstruction algorithm.

ELIGIBILITY:
Inclusion Criteria:

* men and women, aged 18-55 years
* who are able to read and write
* who are able to give voluntary written informed consent
* have no current uncontrolled medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology
* have no history of a neurological or psychiatric disorder, e.g., no DSMIV Axis 1 diagnosis in 2 preceding years, except nicotine dependence in smokers)
* drink less than 21 drinks/week for women and less than 35 drinks per week for men
* have not used marijuana in the past 30 days and have not met criteria for dependence in the past 2 years
* do not suffer from claustrophobia or any MRI contradictions
* nonsmokers (smoked < 40 cigarettes in lifetime with urinary cotinine levels 0-30 ng/mL both at intake evaluation and on scan day)
* smokers (smoked at least 10 cigarettes/day for at least one year with an FTND>3, urine cotinine >150 ng/mL and CO >12 ppm at intake)

Exclusion Criteria:

* psychosis
* presence of acute or unstable medical or neurological illness. Subjects will be excluded from the study if they present with any history of serious medical or neurological illness or if they show signs of a major medical or neurological illness on examination or lab testing including history of seizures, head injury, brain tumor, heart, liver or kidney disease, eating disorder, diabetes.
* regular use of any psychotropic drugs including anxiolytics and antidepressants and other over-the-counter medications and herbal products within the last six months
* pregnancy/breast feeding (as documented by pregnancy testing at screening or on days of the imaging studies),
* suicidal ideation or behavior
* pacemaker or other ferromagnetic material in body.
* use of medications which affect dopamine transmission within 2 weeks of the PET study
* participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits for normal volunteers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cigarette Smokers: Cigarette smokers are subjects who smoke 10 or more cigarettes per day for the past year. All subjects will receive amphetamine at 0.5 kg/mg to induce elevated dopamine levels in the brain. This dosage of amphetamine is given by mouth about 150 minutes prior to the second PET scan.
- Nonsmoking Subjects: Nonsmokers are subjects who have smoked less than 40 cigarettes in their lifetime, and none within the last year. All subjects will receive amphetamine at 0.5 kg/mg to induce elevated dopamine levels in the brain. This dosage of amphetamine is given by mouth about 150 minutes prior to the second PET scan.
Period: Overall Study
Arm/Group | Cigarette Smokers | Nonsmoking Subjects
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cigarette Smokers: Cigarette smokers are subjects who smoke 10 or more cigarettes per day in the past year.
- Nonsmoker Subjects: Nonsmokers are subjects who smoked 40 cigarettes or less in their lifetime, and none within the past year.
- Total: Total of all reporting groups
Arm/Group | Cigarette Smokers | Nonsmoker Subjects | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 3 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 1 | 2
  White, not of Hispanic origin | 4 | 2 | 6
  African American | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Dopamine Levels at Baseline and After Amphetamine Administration as Measured by Percent Change in PET Tracer Binding Potential.
Description: PET images will be obtained in subjects at baseline and after amphetamine administration. Dopamine release will be measured as a percent change in binding potential. Increased dopamine release will result in decreased radiotracer binding because dopamine will displace the radiotracer.
Time Frame: first 90 minute scan at baseline, second 90 minute scan start 150 minutes post amphetamine administration
Measure: Mean (Standard Deviation); unit: percent change in binding potential
Groups:
- Smoking Subjects: Cigarette smokers. These are subjects who smoke at least 10 cigarettes per day for the last year. All subjects will receive amphetamine to induce elevated dopamine levels in the brain at a dose of 0.5mg/kg. They will all receive the amphetamine prior to the second PET scan.
- Nonsmoking Subjects: Nonsmokers. These are subjects who smoked less than 40 cigarettes in their lifetime and none in the last year. All subjects will receive amphetamine to induce elevated dopamine levels in the brain at a dose of 0.5mg/kg. They will all receive the amphetamine prior to the second PET scan
Arm/Group | Smoking Subjects | Nonsmoking Subjects
Number analyzed (Participants) | 6 | 4
percent change in binding potential | -21 (12.0) | -29 (6.3)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Amphetamine: There is only one arm to the study. All subjects will receive amphetamine.
  Amphetamine: All subjects will receive amphetamine to induce elevated dopamine levels in the brain.
Arm/Group | Amphetamine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Preliminary data. Small subject number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No